CLINICAL TRIAL: NCT05311995
Title: Which Trocar Access Site Should We Use in Laparoscopic Appendectomy?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Ersin Gündoğan, Assoc Prof, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021/267
Record Dates: First submitted 2022-03-14; First posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Pain
Keywords: Laparoscopy; Minimally invasive surgery; appendicitis; colorectal
MeSH Terms: conditions — Pain; Appendicitis

STUDY DESIGN:
Intervention Model Description: Four trocar tecnıques groups in literature
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Active Comparator): trocar entry areas:Periumblical, left lower quadrant, suprapubic
  Interventions: Procedure: Only different trocar sites
- Group 2 (Active Comparator): trocar entry areas: Periumblical, left lower quadrant, right lower quadrant
  Interventions: Procedure: Only different trocar sites
- group 3 (Active Comparator): trocar entry areas: Periumblical, right lower quadrant, suprapubic
  Interventions: Procedure: Only different trocar sites
- Group 4 (Active Comparator): trocar entry areas: Periumblical, left lower quadrant, left upper quadrant
  Interventions: Procedure: Only different trocar sites

INTERVENTIONS:
Procedure: Only different trocar sites — Only different trocar sites in literature

SUMMARY:
Open appendectomy has been used in the treatment of appendicitis, which is among the most common emergency pathologies worldwide, since the end of the 19th century. In the 20th century, laparoscopic appendectomy came to the fore and the frequency of use increased gradually. Despite the frequency of laparoscopic appendectomy, there is no consensus on the best way to perform each procedural step. One of these steps is the trocar entry areas. In this study, investigator's aim is to compare the trocar entry areas, which are various reports in the literature, and to find the localization with the optimal usage area. 140 patients who underwent laparoscopic appendectomy between 2021-2022 were randomized into four groups and included in the study. Demographic data, peroperative findings, complications, length of stay and post-operative VAS values of the patients were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent laparoscopic appendectomy

Exclusion Criteria:

patients who underwent open surgery and did not want to be involved in the study process

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-02-20 (Actual)

PRIMARY OUTCOMES:
Pain Intensity measure | 1 year
  self reported pain intensity morning. item is scored 0-10 ( 0: no pain- 10: pain as bad as

CONTACTS AND LOCATIONS:
Locations (1):
- Ersin Gundogan, Kayseri, Kocasinan, Turkey (Türkiye)